CLINICAL TRIAL: NCT02872090
Title: Effects of Long Acting Bronchodilators on CARDiac Autonomic Nervous System Control in Patients With COPD
Brief Title: Effects of Long Acting Bronchodilators on CARDiac Autonomic Control in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: LAB-Card
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P/2015/255
Record Dates: First submitted 2016-08-11; First posted 2016-08-18 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; bronchodilatators; autonomic nervous system; cardiovascular system
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Glycopyrrolate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental): The patients receive once a week during 4 weeks, in the order: indacaterol, tiotropium, glycopyrronium and placebo
  Interventions: Drug: Indacaterol; Drug: Glycopyrronium; Drug: Tiotropium; Drug: Placebo; Procedure: photoplethysmography
- Arm 2 (Experimental): The patients receive once a week during 4 weeks, in the order: tiotropium, glycopyrronium, placebo and indacaterol
  Interventions: Drug: Indacaterol; Drug: Glycopyrronium; Drug: Tiotropium; Drug: Placebo; Procedure: photoplethysmography
- Arm 3 (Experimental): The patients receive once a week during 4 weeks, in the order: glycopyrronium, placebo, indacaterol and tiotropium,
  Interventions: Drug: Indacaterol; Drug: Glycopyrronium; Drug: Tiotropium; Drug: Placebo; Procedure: photoplethysmography
- Arm 4 (Experimental): The patients receive once a week during 4 weeks, in the order: placebo, indacaterol and tiotropium and glycopyrronium
  Interventions: Drug: Indacaterol; Drug: Glycopyrronium; Drug: Tiotropium; Drug: Placebo; Procedure: photoplethysmography

INTERVENTIONS:
Drug: Indacaterol — inhalation
Drug: Glycopyrronium — inhalation
Drug: Tiotropium — inhalation
Drug: Placebo
Procedure: photoplethysmography — inhalation

SUMMARY:
The aim of this interventional, randomized, double-blind, monocentric, cross-over study is to quantify the possible deleterious effect on the cardiac autonomic nervous system control of two long-acting anticholinergic bronchodilatators (tiotropium and glycopyrronium) and one beta-2 agonist long-acting bronchodilatator (indacaterol ) in patients with mild COPD.

DETAILED DESCRIPTION:
This is a cross-over study with randomization in terms of 4 treatments: two long-acting muscarinic antagonists (tiotropium and glycopyrronium), one long-acting beta-adrenoceptor agonist(indacaterol) and placebo.

Each subject will pass 4 experimental random sessions, separated by at least 48 hours given the pharmacokinetic properties of the drugs tested. During each of the 4 sessions, blood pressure will be measured. Drugs inhaled by the patient will be prepared and administered by the nurse according to the randomization schedule. Patients and investigators will be blinded regarding the administered drug/placebo (anonymized inhaler). After 15 minutes (at rest, at neutral temperature), patients will have continuous measurement of blood pressure and heart rate (by a sphygmomanometer) (1) in supine position and (2) after a passive tilt test on a tilt test table.

A flow-volume loop (BDV) will be performed after the tilt table test (measurement of Forced expiratory volume in 1 second (FEV1) and FVC).

ELIGIBILITY:
Inclusion Criteria:

* patients with FEV1 / FVC <70%

Exclusion Criteria:

* beta blocker
* supraventricular rhythm disorder
* previous history of respiratory disease other than COPD
* diabetes
* autonomic dysfunction
* dysautonomia
* renal failure
* long-term oxygen therapy
* history of psychiatric illness

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-03; Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Low-frequency (LF)/High-frequency (HF) ratio in supine position during a tilt table test after bronchodilators inhalation | 10 minutes
  For each patient, the LF/HF ratio after inhalation of an active drug (indacaterol or glycopyrronium or tiotropium) will be compared to LF / HF ratio measured after inhalation of a placebo.

SECONDARY OUTCOMES:
Slope of baroreflex in supine position | 10 minutes
  Drugs vs placebo
LF / HF ratio derived from the spectral analysis of R-R intervals measured after verticalisation during a tilt table test | 10 minutes
  Drugs vs placebo
Total spectral power during a tilt table tes | 20 minutes
  Drugs vs placebo
Value of HF (gross value then normalized according to the average R-R interval) during a tilt table tes | 20 minutes
  Drugs vs placebo
RMSSD (Root Mean Square of the Successive Differences) index during a tilt table test | 20 minutes
  Drugs vs placebo
Variability in blood pressure during a tilt table test | 20 minutes
  Drugs vs placebo

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu VEIL-PICARD, Principal Investigator — CHU Besançon
Locations (1):
- Centre Hospitalier Régional Universitaire, Besançon, France

IPD SHARING:
Plan to Share IPD: No